CLINICAL TRIAL: NCT01870453
Title: Differential Effects of Various Anesthetic Agents on Cognitive Function in Patients With Alzheimer's Disease
Status: Withdrawn | Type: Observational
Why Stopped: Participants recruitment failure
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Zhongcong Xie, Associate Professor of Anaesthesia, Massachusetts General Hospital
Other Study IDs: MassGH-001; HAT-12-237963 (Other Grant/Funding Number: Alzheimer's Association)
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Dementia; Postoperative Care; Cognitive Reserve
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Isoflurane Anesthesia: Recruited subjects that were anesthetized with isoflurane for their surgery.
- Sevoflurane Anesthesia: Recruited subjects that were anesthetized with sevoflurane for their surgery.
- Desflurane Anesthesia: Recruited subjects that were anesthetized with desflurane for their surgery.
- Propofol Anesthesia: Recruited subjects that were anesthetized with propofol for their surgery.

SUMMARY:
The objective of the study is to determine the effects of different anesthetic agents on cognitive function in patients with Alzheimer's disease (AD). The investigators will test the hypothesis that anesthesia with desflurane or propofol, compared to isoflurane or sevoflurane, will have less of an effect on post-operative cognitive dysfunction in patients with AD.

DETAILED DESCRIPTION:
Patients with mild-to-moderate Alzheimer's disease who are scheduled to have elective noncardiac, nonneurologic, nonvascular surgery will be recruited at the Massachusetts General Hospital (MGH). The study will first be introduced to patients at their preoperative surgical clinic appointment by his/her surgeon. If patients are interested in participating, they will notify their surgeons, and subsequent recruitment will take place at the MGH Pre-Admission Testing Area (PATA), a clinic for preoperative evaluation and medical optimization. Patient contact and recruitment, however, will only proceed with permission from (1) the patient him/herself and (2) the patient's surgeon. Per the Partners Human Research Committees-approved criteria, if patients do not have capacity for clinical-decision making but express a willingness to participate in the study, a surrogate (i.e. healthcare proxy and/or family member) co-signature will be required on the consent form. On the day of the subject's surgery, the anesthesia team will be allowed to choose one of four anesthetic options (i.e. propofol anesthesia, isoflurane anesthesia, sevoflurane anesthesia, or desflurane anesthesia) based on clinical preference and appropriateness. The research team will be blinded to the anesthetic to which subjects are assigned. Finally, patients will be followed for one year post-operatively with a battery of cognitive tests to determine differences in cognitive trajectory.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Alzheimer's disease (AD) per Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria.
* Patient recruitment permission granted by his/her surgeon
* Requires general anesthesia for elective noncardiac, nonneurologic, nonvascular surgery.

Exclusion Criteria:

* History of neurologic or psychiatric disease (i.e. stroke, psychosis, etc.)
* Non-native English speaker
* Severe visual or auditory disorder
* Sensitivity to sulfites (some propofol formulations at MGH may contain sodium metasulfite).
* Asthma (sulfite sensitivity is seen more frequently in asthmatic than in non-asthmatic people).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 100 study participants with mild-to-moderate AD who are scheduled to have elective noncardiac, nonneurologic, nonvascular surgery will be recruited at MGH. Surgeons will first introduce the study to patients at their preoperative surgical clinic visit. If a patient expresses interest in the study, and with permission of the surgeon, the patient will then be contacted by study staff at his/her PATA preoperative evaluation and medical optimization clinic visit. Recruitment, screening, and enrollment will then occur at the patient's PATA clinic visit.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-10 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function | 1 week pre-operatively to 1 year post-operatively
  Cognitive function will be assessed using a battery of neuropsychological tests in the domains of attention and executive functions (Trail Making Test, Verbal Fluency Test, Category Switching Test, Symbol Digit Modalities Test), memory (Hopkins Verbal Learning Test-R, Brief Visual Memory Test-R), visuospatial functions (Benton Judgement of Line Orientation Test), and language (Category Fluency Test).

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States